CLINICAL TRIAL: NCT06606379
Title: Impact of Different Separation Methods on Proximal Contact Tightness and Contour of Compound Class ii Nanohybrid Resin Composite Restorations: Randomized Clinical Trial
Brief Title: Impact of Different Separation Methods on Proximal Contact Tightness and Contour of Compound Class ii
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hadeer Hesham Mohamed, Dr. Hadeer Hesham, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IMPACT OF SEPARATION METHODS
Record Dates: First submitted 2024-09-18; First posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Proximal Caries
MeSH Terms: interventions — Methods

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- C (comparator) (Active Comparator): Nickel titanium 3D-fusion ring (Garrison, USA)
  Interventions: Device: C (comparator)
- I1 (Intervention) (Experimental): Resin ring (DR- Resin ring, Egypt)
  Interventions: Device: I1 (Intervention)
- I2 (Intervention) (Experimental): Elliot separator (Pfingst & Co, South Plainfield, NJ, USA)
  Interventions: Device: I2 (Intervention)
- I3 (Intervention) (Experimental): Stainless Steel Metal ring (TOR VM ring, Moscow, Russia)
  Interventions: Device: I3 (Intervention)

INTERVENTIONS:
Device: I1 (Intervention) — Resin ring (DR- Resin ring, Egypt)
  Arms: I1 (Intervention)
Device: I2 (Intervention) — Elliot separator (Pfingst & Co, South Plainfield, NJ, USA)
  Arms: I2 (Intervention)
Device: I3 (Intervention) — Stainless Steel Metal ring (TOR VM ring, Moscow, Russia)
  Arms: I3 (Intervention)
Device: C (comparator) — Nickel titanium 3D-fusion ring (Garrison, USA)
  Arms: C (comparator)

SUMMARY:
The aim of this study is to evaluate the interdental separation of various separation systems and their impact on the proximal contact tightness and contour in compound class II nanohybrid resin composite restorations.

DETAILED DESCRIPTION:
The target population consists of adult patients aged 25-40, with posterior compound proximal carious cavities (ICDS score 4 or 5) in molars. The interventions under investigation include three different separation systems: the Resin ring (DR-Resin ring, Egypt), Elliot separator (Pfingst & Co, USA), and Stainless Steel Metal ring (TOR VM ring, Russia). These systems will be compared to a Nickel titanium 3D-fusion ring (Garrison, USA). The primary outcomes assessed are proximal contact tightness and form/contour, measured visually according to FDI criteria, with scoring systems adapted from Hickel et al. (2023). Secondary outcomes, such as patient comfort (measured by a pain rating scale), and the emergence profile (assessed via bitewing radiographs), will also be considered. Data will be collected immediately postoperatively (T0), at 30 days (T1), and after 6 months (T2). The study will be conducted as a randomized clinical trial. The null hypothesis suggests that there will be no significant differences in proximal contact tightness or contour across the different separation systems used.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals with posterior compound proximal carious cavities in molars.
2. Age of (25-40) years.
3. Molars with compound proximal carious cavities score 4 or 5 ICDS.
4. Vital upper or lower posterior teeth with no signs of irreversible pulpitis.
5. Presence of adjacent and opposing teeth with normal occlusion

Exclusion Criteria:

1. Patients with major systemic disorders or xerostomia.
2. Patients with periodontal disease.
3. Patients with para-functional habits.
4. Presence of malocclusion or signs of pathological teeth wear
5. Non vital teeth or teeth with signs of pulpal pathology.
6. Teeth mobility or clinical attachment loss.

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Proximal Contact tightness (Success rate) | From enrollment to the end of treatment at 6 months
  Visual examination and 25-/50-/100-µm blade according to FDI Criteria

SECONDARY OUTCOMES:
Form and Contour | From enrollment to the end of treatment at 6 months
  Visual examination according to FDI Criteria
Patient Comfort | From enrollment to the end of treatment at 6 months
  Pain rating scale
Emergence profile | From enrollment to the end of treatment at 6 months
  Bitewing Radiographs

CONTACTS AND LOCATIONS:
Overall Officials: Hadeer H Mohamed, MSC. degree, Principal Investigator — Assistant Lecturer of Conservative Dentistry, Faculty of Dentistry Cairo University, Egypt.

IPD SHARING:
Plan to Share IPD: Undecided